CLINICAL TRIAL: NCT05032404
Title: BNT 103 Usability and User Engagement
Brief Title: Blue Note Therapeutics Product BNT 103 Usability and User Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blue Note Therapeutics (Industry)
Collaborators: Healthcare Innovation Technology Lab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PROT002 - Test Plan 01 Rev A
Record Dates: First submitted 2021-08-31; First posted 2021-09-02 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- BNT103 (Experimental): All participants receive BNT103. BNT103 provides 10 sessions over approximately 10 weeks.
  Interventions: Device: BNT103

INTERVENTIONS:
Device: BNT103 — BNT-103™ is a prescription digital therapeutic specifically designed to treat the symptoms of anxiety and depression related to cancer. There are 10 sessions provided over approximately 10 weeks.

SUMMARY:
This test aims to explore product development-focused usability and user engagement.

DETAILED DESCRIPTION:
Sponsor is testing an innovative peer-to-peer communication tool during this trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient can read, write, and speak in English
* Patient is between the ages of 35-55
* Diagnosed with Stage I-III breast cancer
* In active treatment or within 3 months of ending active treatment and under the care of a clinician at time of study
* Apple mobile phone or tablet user
* Willing to participate in study protocol

Exclusion Criteria:

* Any participant not meeting inclusion criteria

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Diagnosed with breast cancer
Enrollment: 15 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Mean mHealth App Usability Questionnaire (MAUQ) for Standalone mHealth Apps Used by Patients | Baseline up to Week 7
  Higher scores indicate higher ease of use / easier to use applications

SECONDARY OUTCOMES:
Measure of Current Status - Anxiety (MOCS-A) | Baseline up to Week 7
  The MOCS-A is a 13-item self-report measure developed to assess participants' current self-perceived status on: the ability to relax at will, recognize stress-inducing situations, restructure maladaptive thoughts, be assertive about needs, and choose appropriate coping responses as needed, higher scores indicate greater self-perceived proficiency with these skills.

CONTACTS AND LOCATIONS:
Overall Officials: Dianne Shumay, PhD, Principal Investigator — Blue Note Therapeutics, Inc
Locations (1):
- Blue Note Therapeutics, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antoni MH, Lechner S, Diaz A, Vargas S, Holley H, Phillips K, McGregor B, Carver CS, Blomberg B. Cognitive behavioral stress management effects on psychosocial and physiological adaptation in women undergoing treatment for breast cancer. Brain Behav Immun. 2009 Jul;23(5):580-91. doi: 10.1016/j.bbi.2008.09.005. Epub 2008 Sep 20. PMID 18835434